CLINICAL TRIAL: NCT03997604
Title: A Descriptive, Prospective Clinical Study to Evaluate Fit and Quality of Full Dentures Fabricated by Additive Manufacturing
Brief Title: A Descriptive, Prospective Clinical Study to Evaluate Full Dentures Fabricated by Additive Manufacturing
Status: Withdrawn | Type: Observational
Why Stopped: The Dental service organization that the Sponsor was working with did not meet the Sponsor's internal requirements for performing the clinical trial. As a result the study was withdrawn without any participant enrollment.
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Other Study IDs: PRPA2290/CR-01
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Full Dentures created by additive manufacturing — Full dentures created by Additive manufacturing (Carbon Printers)
  Other Names: Lucitone 3D print resin dentures

SUMMARY:
This investigation is undertaken to evaluate the workflow and concomitant products to create full dentures by using Additive Manufacturing (AM) technology, i.e. Digital Light Processing™ Technology (Carbon 3D) to restore fully edentulous jaws. The assessment includes quality of materials provided by Dentsply Sirona Lab by using printers for Additive Manufacturing (M2 series, Carbon 3D 1089 Mills Way, Redwood City, CA 94063). This assessment will be done by clinical review of the AM dentures on fit and quality. In addition, the trial includes a patient survey to assess current dentures and the new AM dentures with a subjective comparison of both.

DETAILED DESCRIPTION:
Study Design:

* This descriptive, prospective, clinical investigation will be conducted on approximately forty (40) enrolled subjects at four (4) sites in the US.
* Treatment of subjects encompasses all steps to fabricate new dentures for maxilla and mandible (no greater than five (5) visits; 30-60 min. chair time per appointment).
* The subjects will be followed 7-10 days after final delivery of the denture for function check.
* Long-term follow-up will be performed after 6 months, 12 months, 24 months and 36 months to assess fit, function, and esthetics under function performed by the dental professional and by capturing according feedback by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Subject has given written consent to participate in the trial.
* Subject is in good general health.
* Subject requires a new removable full denture for both jaws.
* Subject is completely edentulous in the maxilla and mandible.
* Subject is already wearing a full denture in the maxilla and mandible.
* Subject is willing to undergo dental treatment to receive a new full denture for both jaws.
* Subject confirms availability for treatment and all indicated follow-up visits.

Exclusion Criteria:

* Subject is younger than 18 years.
* Subject is pregnant.
* Subject has disabilities that do not allow a regular dental treatment.
* Subject with some systemic medical complications that cause difficulty in impression taking or judging occlusion of device.
* Subject is currently participating in another study.
* Subject has an allergic history regarding materials used in this trial.
* Subject with xerostomia/ dry-mouth syndrome.
* Lack of compliance is expected.
* Those subjects who cannot provide informed consent for any reason
* Acute stomatitis.
* Status after tumor treatment in head-neck region (removal, radiotherapy).
* Acute cancer.
* Incomplete hard and/or sift tissue in the oral cavity.
* Muscle and/or nerve damage in the head-neck region.
* Insufficient vertical height and/or insufficient mouth opening.
* Resilient hyperplastic mucosa ("flappy ridges").
* Bruxism.
* Insufficient oral hygiene. The existing dentures should have no visible calculus.
* Previously enrolled in the present investigation.
* Involvement in the planning and conduct of the clinical investigation. (applies to all Dentsply Sirona & Carbon 3D staff, investigational site staff/Affordable staff and third party vendor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigational device is part of a treatment concept for edentulous patients of all ages, gender and races. The incidence for tooth loss has not declined over years, and the prevalence for edentulism is significantly higher for adults 50 years and older15, 16. For this descriptive two-part survey, no minimum number of patients is defined, but to achieve a reasonable subject number, a minimum of forty (40) patients will be enrolled, i.e. 80 dentures will be fabricated within this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-10-29 (Estimated); Study Completion 2022-10-29 (Estimated)

PRIMARY OUTCOMES:
assessment of the fit of the denture | 7 days after final placement of dentures
  Assessment of the fit of the new dentures in comparison to the previous prostheses in the mouth immediately after first insertion by dentist. A questionnaire of Assessment of fit by ranking from
  * Much worse
  * Worse
  * Same
  * Better
  * Much better

SECONDARY OUTCOMES:
Aesthetics of dentures | 7 days after final placement of dentures
  patients overall satisfactions of the dentures aesthetics. A questionnaire of assessment of fit by ranking from
  * Much worse
  * Worse
  * Same
  * Better
  * Much better
Function of dentures | 7 days after final placement of dentures
  patients overall satisfaction of dentures to masticate. Assessment of fit by ranking from
  * Much worse
  * Worse
  * Same
  * Better
  * Much better
Patient's satisfaction with denture and treatment | 36 months after final placement
  Patients are asked to compare existing and new denture by using a survey. a Questionnaire Assessment of fit by ranking from
  * Much worse
  * Worse
  * Same
  * Better
  * Much better
Dentist's satisfaction with treatment | 7 Days after final placement
  Assessment of treatment process in comparison to traditional denture fabrication process. A questionnaire Assessment of fit by ranking from
  * Much worse
  * Worse
  * Same
  * Better
  * Much better
Health of oral cavity and related tissues | 36 months after final placement
  Continuously clinical intra-oral inspection of oral landmarks and tissues with regard to any findings. ** *parameters according to Grandmont, ** Scottish Dental effectiveness program. Assessment of by scoring:
  * pigmented
  * ulcus
  * white
  * red
  * swelling
  * negative

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Affordable Dentures and Implants, Northglenn, Colorado
  - Wagner Denture Group 801 Encino Pl NE A3, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celebic A, Knezovic-Zlataric D, Papic M, Carek V, Baucic I, Stipetic J. Factors related to patient satisfaction with complete denture therapy. J Gerontol A Biol Sci Med Sci. 2003 Oct;58(10):M948-53. doi: 10.1093/gerona/58.10.m948. PMID 14570864
- [Background] Schwindling FS, Bomicke W, Hassel AJ, Rammelsberg P, Stober T. Randomized clinical evaluation of a light-cured base material for complete dentures. Clin Oral Investig. 2014;18(5):1457-65. doi: 10.1007/s00784-013-1110-4. Epub 2013 Sep 21. PMID 24057919